CLINICAL TRIAL: NCT03413813
Title: Prospective Observational Registry of Patients With a Bioabsorbable Magnesium Stent Implant -MAGMARIS- in Usual Clinical Practice
Brief Title: Registry of Patients With a Bioabsorbable Magnesium Stent Implant MAGMARIS in Usual Clinical Practice
Acronym: MAGMARIS
Status: Completed | Type: Observational
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Andres Iñiguez Romo, MD, Head of cardiology, Spanish Society of Cardiology
Other Study IDs: MAGMARIS-ES
Record Dates: First submitted 2017-12-21; First posted 2018-01-29 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease
Keywords: Magmaris
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Magmaris — Severe stenosis de novo, in native coronary arteries, treated with percutaneous coronary intervention with scaffold implantation.
  Other Names: Bioresorbable scaffold

SUMMARY:
The safety and efficacy of percutaneous coronary revascularization has been progressively increasing since its inception, and the problem of restenosis has been minimized.

The efficacy and safety data of the Magmaris stent are quite high, in selected cases.

The objective is to evaluate the efficacy and safety of the bioabsorbable stent MAGMARIS in the percutaneous treatment of severe coronary disease (in vessels between 2.7mm and 3.75 mm) in routine clinical practice in poorly selected populations.

DETAILED DESCRIPTION:
This is a multicentre, observational, prospective registry of patients without a control group designed to evaluate the efficacy and safety of the bioabsorbable coronary device, according to the indications for use, in routine clinical practice in a consecutive number of patients undergoing percutaneous coronary intervention (PCI) in de novo coronary arteries lesions in a native coronary artery.

After the implantation of the device, a telephone or face-to-face follow-up will be carried out in the first month, at 12 months and at 24 months.

A total of 445 patients are expected to be included in the registry. Patients, will be included consecutively in each center over a year. A selection period of 23 months or until the estimated sample size has been planned, with a follow-up of two years. Subsequently, it will take at least 3 months for data analysis, another 2 months for the final report and at least 3 more months for the publication of the results for publication. This implies that the total duration of the study will be 55 months counted from the inclusion of the first patient.

The procedure will be carried out according to the usual practice of each center, paying special attention to the correct expansion of the scaffold, postdilating with non-compliant balloons when necessary.

The collection of information from the study will be carried out on a data collection template in electronic format, which will include clinical, anatomical, procedural and follow-up data; in baseline circumstances, during hospitalization, after discharge and throughout follow-up at 1, 12, and 24 months. The source documents will be the patient's medical records collected at the center.

The monitoring will be done monthly and online. Two face-to-face monitoring will be done to 20% of the patients, during the inclusion and follow-up phases. Afterwards, a face-to-face monitoring will be carried out for the closing visit.

Descriptive and univariate statistics will be performed. The primary variable is the MACE rate at 12 months, composed of cardiac death, myocardial infarction and TLR induced by ischemia (primary objectives). The secondary variables will be combined indices of events both in the hospital phase, and after discharge in the follow-up at 1, 12 and 24 months.

A final report will be prepared containing all the results of the study, in a period of 6 months once the same one finalized. The participating researchers and the Ethical Committees of the hospitals will be informed about this.

ELIGIBILITY:
Inclusion Criteria:

* BASIC CRITERIA:

  * Patients who agree to participate in the study, signing the informed consent form.
  * The implantation of the bioresorbable MAGMARIS coronary device used according to the indications for use in the center's routine clinical practice.
  * Patients of both sexes over 18 years of age.
  * The patient does not present any contraindication regarding the taking of dual therapy of antiplatelet therapy with aspirin indefinitely and with thienopyridines for at least the first 6 months.
* CLINICAL CRITERIA:

  * Angor stable or anginal equivalent diagnosis of stable chronic ischemic heart disease.
  * Documented silent ischemia
  * Acute coronary syndrome (excluding AMI with ST-segment elevation <24 hours)
  * Angina Equivalent
* ANGIOGRAPHICAL CRITERIA:

  * One or more de novo lesions (stenosis> 70% by visual estimation or> 50% by estimation of quantitative automatic angiography) in native coronary arteries.
  * Vessel reference diameter ≥2.7 and ˂3.75.
  * Maximum length of the lesion to be treated must be less than the nominal length of the device (15 mm, 20 mm, 25 mm) or capable of being covered with more than one scaffold implanted in an overlapped manner by at least 1 mm with respect to the adjacent.

Exclusion Criteria:

* CLINICS:

  * Cardiogenic shock
  * Acute Myocardial Infarction (first 24 hours).
  * Concurrent diseases with life expectancy of less than 1 year
  * Women of reproductive age who do not use contraception.
  * Women who are pregnant or breast-feeding.
  * Allergies: AAS, Thienopyridines, Magnesium.
* ANATOMICS:

  * Main coronary artery lesion
  * Lesion in aorto-coronary graft of saphenous vein or mammary artery.
  * Intra-stent restenosis lesion.
  * Lesion chronic total occlusion.
  * Bifurcation lesion
  * Severely calcified or severely tortuous coronary artery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease by de novo lesions in native coronary arteries, candidates for revascularization with coronary stent.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
A combined rate (incidence of events) of: | 12 months
  The cardiac death (incidence of events).
A combined rate (incidence of events) of: | 12 months
  Myocardial infarction (incidence of events)
A combined rate (incidence of events) of: | 12 months
  Revascularization of the treated lesion (TLR) induced by ischemia (incidence of events)

SECONDARY OUTCOMES:
The event rate will be calculated for: | 24 months
  Cardiovascular deaths
The event rate will be calculated for: | 24 months
  Non-cardiovascular deaths
The event rate will be calculated for: | 24 months
  Myocardial infarctions (MI: QMI and NQMI, TV, NTV)
The event rate will be calculated for: | 24 months
  Revascularization of the treated lesions induced by ischemia (ID-TLR)
The event rate will be calculated for: | 24 months
  Revascularization of the treated vessels induced by ischemia (ID-TVR)
The event rate will be calculated for: | 24 months
  All revascularizations (PCI vs. CABG)
The event rate will be calculated for: | 24 months
  Thrombosis of the device. Classification (acute, sub-acute, delayed) and evidence classification (definitive, probable, possible)
The event rate will be calculated for: | 24 months
  Overlapping devices and features
The event rate will be calculated for: | 24 months
  The immediate success of the device
The event rate will be calculated for: | 24 months
  The immediate success if the procedure
The event rate will be calculated for: | 24 months
  The failure of the lesion treated through a combined rate of cardiac death, TV-IM and ID-TLR: (Failure of treated lesion (TLF))
The event rate will be calculated for: | 24 months
  The failure of the vessel treated through a combined rate of cardiac death, total myocardial infarction and ID-TVR: (Failure of treated vessel (TVF))
The rate of: | 24 months
  Overlapping stents will be calculated in relation to those implanted, and the relation with the appearance of clinical events.
The rate of: | 24 months
  Image parameters will be calculated in the cases in which, in the opinion of the researcher, coronary function or intravascular imaging tests have been performed (FFR, IVUS, OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Andres I Romo, MD, PhD, Study Director — Spanish Society of Cardiology
Locations (31):
- Spain (31):
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario General de Castellón, Castellon, Castellón
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario Clinic de Barcelona, Barcelona
  - Hospital Universitario Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital Universitario General de Ciudad Real, Ciudad Real
  - Hospital Universitario Doctor Josep Trueta, Girona
  - Hospital San Cecilio-Campus de la Salud, Granada
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Clínico de Valencia, Valencia
  - Hospital Universitario General de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario de Áraba, Vitoria-Gasteiz, Álava